CLINICAL TRIAL: NCT01311882
Title: A Multiple Dose Study to Evaluate Next Day Effects of MK-4305 on Driving Performance in Healthy Non-Elderly Subjects
Brief Title: A Study to Evaluate Next Day Effects of MK-4305 on Driving Performance (MK-4305-035 AM1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 4305-035
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — suvorexant; zopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- MK-4305 40 mg (Experimental): Day 1 and Day 8- 4 x 10 mg MK-4305 and 1 x 7.5 mg zopiclone grossly matching placebo; Days 2-7 - 4 x 10 mg MK-4305
  Interventions: Drug: MK-4305 40 mg; Drug: Grossly Matching Placebo for Zopiclone
- MK-4305 20 mg (Experimental): Day 1 and Day 8- 2 x 10 mg MK-4305 and 2 x 10 mg MK-4305 matching placebo and 1 x 7.5 mg zopiclone grossly matching placebo; Days 2-7 - 2 x 10 mg MK-4305 and 2 x 10 mg MK-4305 matching placebo
  Interventions: Drug: MK-4305 20 mg; Drug: Grossly Matching Placebo for Zopiclone; Drug: Matching Placebo for MK-4305
- Zopiclone 7.5 mg (Active Comparator): Day 1 and Day 8- 1 x 7.5 mg zopiclone and 4 x 10 mg MK-4305 matching placebo; Days 2-7- 4 x 10 mg MK-4305 matching placebo
  Interventions: Drug: Zopiclone; Drug: Matching Placebo for MK-4305
- Placebo (Placebo Comparator): Day 1 and Day 8- 4 x 10 mg MK-4305 matching placebo and 1 x 7.5 mg zopiclone grossly matching placebo; Days 2-7 - 4 x 10 mg MK-4305 matching placebo
  Interventions: Drug: Grossly Matching Placebo for Zopiclone; Drug: Matching Placebo for MK-4305

INTERVENTIONS:
Drug: MK-4305 40 mg — 4 x 10 mg MK-4305 tablets
  Arms: MK-4305 40 mg
Drug: MK-4305 20 mg — 2 x 10 mg MK-4305 tablets
  Arms: MK-4305 20 mg
Drug: Zopiclone — 1 x 7.5 mg Zopiclone tablet
  Other Names: Zimovane
  Arms: Zopiclone 7.5 mg
Drug: Grossly Matching Placebo for Zopiclone — Grossly Matching Placebo for Zopiclone
  Arms: MK-4305 20 mg; MK-4305 40 mg; Placebo
Drug: Matching Placebo for MK-4305 — Matching Placebo for MK-4305
  Arms: MK-4305 20 mg; Placebo; Zopiclone 7.5 mg

SUMMARY:
This is a study to evaluate next-day residual effects of MK-4305 on highway driving performance in healthy, non-elderly participants.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of reproductive potential must agree to use (and/or have their partner use) acceptable methods of birth control beginning at least 2 weeks prior to the administration of the first dose of study drug throughout the study
* Has a body mass index (BMI) within the range of 18 to 30 kg/m^2
* Possesses a valid driver's license for 3 years or more with at least 5000 km/year on average within the last 3 years
* Is capable of driving a manual transmission vehicle and is willing to drive on a highway
* Is judged to be in good health
* Has a regular sleep pattern
* Is not visually impaired

Exclusion Criteria:

* Has a history of a persistent sleep abnormality
* Has neurological disease/cognitive impairment
* Has a history of cataplexy
* Is a regular user of sedative-hypnotic agents
* Is allergic to zopiclone
* Has traveled across 3 or more time zones (transmeridian travel) in the last 2 weeks prior to study start and will travel across 3 or more time zones throughout study duration
* Works a night shift and is not able to avoid night shift work within 1 week before each treatment visit
* Is pregnant or nursing
* Does not qualify as a proficient driver according to the driving instructors evaluation of subject's driving on the driving test practice session

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Mean differences of standard deviation of lateral position (SDLP) on highway driving between MK-4305 and placebo | Day 2

SECONDARY OUTCOMES:
Mean differences of standard deviation of lateral position (SDLP) on highway driving between zopiclone and placebo | Day 2
Mean differences of standard deviation of lateral position (SDLP) on highway driving between MK-4305 and placebo | Day 9
Mean differences of standard deviation of lateral position (SDLP) on highway driving between zopiclone and placebo | Day 9
Mean standard deviation of speed (SDS) on highway driving (MK-4305 versus placebo) | Day 2 and Day 9
Word learning test (MK-4305 versus placebo) | Day 2 and Day 9
Body sway area: Area of the 95% confidence ellipse enclosing the center of pressure (A95) (MK-4305 versus placebo) | Day 2 and Day 9
Number of participants with adverse events | Up to 14 days after last dose
Number of participants discontinued from study due to adverse events | Up to 14 days after last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Merck Sharp & Dohme B.V., Haarlem, Netherlands

REFERENCES:
- [Background] Vermeeren A, Sun H, Vuurman EF, Jongen S, Van Leeuwen CJ, Van Oers AC, Palcza J, Li X, Laethem T, Heirman I, Bautmans A, Troyer MD, Wrishko R, McCrea J. On-the-Road Driving Performance the Morning after Bedtime Use of Suvorexant 20 and 40 mg: A Study in Non-Elderly Healthy Volunteers. Sleep. 2015 Nov 1;38(11):1803-13. doi: 10.5665/sleep.5168. PMID 26039969